CLINICAL TRIAL: NCT04808154
Title: A Phase I Single Dose Study to Investigate the Safety, Tolerability and Pharmacokinetic Profile of SNP-630 in Health Subjects.
Brief Title: A Phase I Study to Investigate the Safety, Tolerability and Pharmacokinetic Profile of SNP-630 in Health Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sinew Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNP-630-101
Record Dates: First submitted 2021-02-09; First posted 2021-03-22 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: SNP-630
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- test drug (Experimental): Powder for oral solution of SNP-630.
  Interventions: Drug: SNP-630

INTERVENTIONS:
Drug: SNP-630 — Subjects will receive one single dose of SNP-630 at Day 1. Blood and urine samples will be obtained to determine the PK of orally administered SNP-630.

SUMMARY:
To evaluate the safety, tolerability and Pharmacokinetic profile of SNP-630 when oral administered to healthy subjects.

DETAILED DESCRIPTION:
A Phase 1 Single Dose Study to investigate the safety, tolerability and Pharmacokinetic profile of SNP-630 in Health Subjects To evaluate the safety, tolerability and Pharmacokinetic profile of SNP-630 when oral administered to healthy subjects.

This is a phase 1, open-label, single-dose study to assess its safety, tolerability and pharmacokinetic profile of SNP-630 in 14 health volunteers. Subjects will receive oral SNP-630 at a dose of 720 mg to assess its safety, tolerability and pharmacokinetic profile.

After written informed consent has been obtained, all screening procedures and tests that establish study eligibility will be performed within 28 days prior to day -1 visit.

The primary endpoint is to assess the following variable:

Clinical safety observations will include Adverse Events (AEs), vital sign measurements, 12-lead ECG and clinical laboratory assessments. Safety data will be tabulated and where appropriate, analyzed by the use of descriptive statistics. Safety data will be tabulated by system organ class and preferred term and will be further classified by relationship to treatment. The probability of safety events will be estimated and with associated 95% corresponding confidence intervals for each cohort using the binomial distribution.

Participants are free to withdraw from participation in the study at any time upon request

ELIGIBILITY:
Inclusion Criteria:

* A subject can participate in the study only if all the following criteria are met:

  1. Between 20 and 45 years
  2. Body weight 55 - 95 kg and body mass index (BMI) within the range 19 - 30 kg/m2
  3. Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests, vital signs and 12-lead ECG. (A subject with a clinically insignificant abnormality or laboratory parameter(s) may be included only if the Investigator documents that the finding is unlikely to represent a safety risk and will not interfere with the study procedures.)
  4. Male or Female of non-reproductive potential
  5. Able to provide written informed consent, and understand and comply with the requirements of the study

     Exclusion Criteria:
* Subjects who meet any of the following criteria are not eligible to enter the study:

  1. History of any significant medical condition (e.g. Cardiovascular, pulmonary, metabolic, renal, gastrointestinal, urological, psychological disease, etc.)
  2. With any surgical or medical condition possibly affecting drug absorption (e.g. cholecystectomy, gastrectomy, bowel disease, etc.), distribution, metabolism or excretion
  3. History of liver disease, or known hepatic or biliary abnormalities
  4. Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test (anti-HBc Ab) result at screening
  5. AST, ALT, gamma-GT and total bilirubin >1.0x ULN
  6. Creatinine >1.0 x ULN
  7. Donation of blood or blood products in excess of 500 mL within 3 months
  8. Has participated in a clinical trial and has received an investigational product within 3 months prior to dosing
  9. Pregnant or lactating
  10. Anticipated requirement for any prescription medication during the study.
  11. History of sensitivity to any of the study medications, or components thereof or a history of anaphylaxis or severe allergy to drug or other substances
  12. History or presence of alcohol abuse, defined as consumption of more than 210 mL of alcohol per week (the equivalent of 14 glasses of 120-mL wine or 14 cans of 350-mL beer), or other substance abuse within the prior two years

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs): | 6 days
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

SECONDARY OUTCOMES:
Pharmacokinetic profile of SNP-630 | 6 days
  Concentrations of SNP-630 and it metabolites in plasma and urine will be measured by a specific and sensitive LC/MS/MS method developed in the laboratory of Clinical Pharmacokinetic Laboratory of Tri-Service General Hospital. According to the pharmacokinetic parameters of SNP-630 and its metabolites in health subjects oral SNP-630 to assess the safety information.The study will be conducted to validate the precision, accuracy (including with-run and between-run variation), linearity, specificity, reproducibility, limit of quantitation based on recovery studies. Assays will be performed in the laboratory of Clinical Pharmacokinetic Laboratory of Tri-Service General Hospital. Spiked samples of known concentrations will be analyzed together for quality control of the assay method.

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No